CLINICAL TRIAL: NCT05371743
Title: Plasma microRNA Levels and Some Cytokines Expression in Patients With Primary Immune Thrombocytopenic Purpura (ITP)
Brief Title: Plasma microRNA Levels and Some Cytokines Expression in Patients With ITP Primary Immune Thrombocytopenic Purpura (ITP)
Acronym: microRNAITP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Noha Saber Shafik, lecturer of Medical Microbiology and Immunology, faculty of medicine, Sohag University
Other Study IDs: 290-2022
Record Dates: First submitted 2022-05-07; First posted 2022-05-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: MicroRNA, ITP, IL17
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — After informed patient consent, Blood samples will be taken when patients visited the hospital and an ITP diagnosis was made. For persistent, chronic, and acute ITP patients.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ITP patients: Patients will be recruited from the internal department- hematology unit outpatient clinic of El Minia University Hospital in collaboration with the clinical pathology department of El Minia University Hospital and the biochemistry department of Minia and Sohag University. Exclusion criteria:
  1. Secondary causes of ITP as systemic lupus erythematous (SLE), viral infections (HIV, hepatitis B or C infections)
  2. Other underlying medical diseases that may cause thrombocytopenia as:
     * malignancy
     * megaloblastic anemia
     * aplastic anemia
     * lymphoproliferative disorders
     * liver disease
     * renal impairment
     * pregnancy
  3. Organomegally and/or lymphadenopathy.
  4. Recent history of vaccination.
  5. Recent evidence of bacterial infection.
  Interventions: Diagnostic Test: Plasma RNA isolation, qPCR analysis of micro RNA; Diagnostic Test: estimation of serum level of IL2; Diagnostic Test: estimation of serum level of IL17
- normal individuals: Blood samples will be taken from normal individuals.

INTERVENTIONS:
Diagnostic Test: Plasma RNA isolation, qPCR analysis of micro RNA — qPCR will be performed using Taqman microRNA assays (Applied Biosystems, Foster City, CA, USA) according to the manufacturer's protocol. Total RNAs going to be used to make cDNAs using TaqMan microRNA RT Kit. Diluted cDNAs were mixed with TaqMan Universal PCR Master Mix (No AmpErase UNG). Taqman miRNA assay will run in the 7500 Real-Time PCR System (Applied Biosystems). miR-39 also will be used as an exogenous control. All assays will be done in triplicates. The expression levels will be evaluated using the comparative cycle threshold (∆∆_Ct) method
  Groups: ITP patients
Diagnostic Test: estimation of serum level of IL2 — 2ml of patient serum will be used to measure IL 2 in patients with different groups by ELISA technique.
  The techniques will be done in the central research laboratory in Sohag university hospital
  Groups: ITP patients
Diagnostic Test: estimation of serum level of IL17 — 2ml of patient serum will be used to measure IL17 in patients with different groups by ELISA technique.
  The techniques will be done in the central research laboratory in Sohag university hospital
  Groups: ITP patients

SUMMARY:
Immune thrombocytopenia (ITP) is an autoimmune disease characterized by low platelet counts with or without mucocutaneous bleeding (McMillan, 2007). Like the majority of autoimmune diseases, ITP is an organ-specific disease, and abnormalities in the regulation of the immune system have been shown to play an important role in the initiation and/or perpetuation of the disease (McKenzie et al.,2013).

Still, immune thrombocytopenia (ITP) is a significant clinical problem due to chronicity, treatment cost, occurrence mainly in, young, and relatively poorer quality of life

DETAILED DESCRIPTION:
In recent years the critical role of miRNAs has been established in many diseases, including autoimmune disorders. Immune thrombocytopenic purpura (ITP) is a predominant autoimmune disease, in which aberrant expression of miRNAs has been observed, suggesting that miRNAs are involved in its development (Jafarzadeh et al., 2021). Studies have also shown that cell-free miRNAs in circulation are stable and that such miRNAs may be exploited as novel disease markers (Etheridge et al.,2011) and ( van Rooij et al., 2008).

MicroRNAs (miRNAs) are endogenous small RNAs, usually 18-25 nucleotides in length. These non-coding RNAs regulate gene expression by several mechanisms, such as repressing protein translation and altering mRNA stability (Ambros, 2008. Bartel,2004). In humans, >2,000 miRNAs have been discovered. The functional significance of the majority of the identified miRNAs has yet to be fully elucidated. Studies have shown that miRNAs play important roles in hematopoietic differentiation, e. g. megakaryocytopoiesis. (Garzon et al., 2008) and erythropoiesis ( Masaki et al., 2007 )and (Bruchovaetal., 2007), and in hematological malignancies (Rossi et al.,2010) and (Visone et al.,2009). More recently, miRNAs have also been implicated in cellular immune responses that contribute to ITP (Jernas et al., 2013) and (McKenzie etal., 2013). It was found that 23 differentially expressed miRNAs in ITP (14 up-regulated and 9 down-regulated) Altered miRNA expression may occur in specific diseases and at specific disease stages (Martin et al., 2012) Also, Recent studies have demonstrated that Th17, which is characterized for its production of IL-17, is elevated in ITP patients (Hu et al., 2012) and (Huber et al., 2007). IL-17 belongs to the IL-17 cytokine family. Increased IL-17 expression has been observed in various autoimmune diseases, such as rheumatoid arthritis (RA) ( Roeleveld et al., 2013) and systemic lupus erythematosus (SLE) (Ballantine et al., 2014). This evidence suggests that IL-17 may be associated with autoimmune diseases.

ELIGIBILITY:
Inclusion Criteria:

* ITP patients

Exclusion Criteria:

* 1- Secondary causes of ITP as systemic lupus erythematosus (SLE), viral infections (HIV, hepatitis B or C infections) 2- Other underlying medical diseases that may cause thrombocytopenia as:
* malignancy
* megaloblastic anemia
* aplastic anemia
* lymphoproliferative disorders
* liver disease
* renal impairment
* pregnancy 3-Organomegally and/or lymphadenopathy. 4-Recent history of vaccination. 5-Recent evidence of bacterial infection.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This is a cross-sectional study. Patients will be recruited from the internal department- hematology unit outpatient clinic of El Minia University Hospital in collaboration with the clinical pathology department El Minia University Hospital and the biochemistry department of Minia and Sohag University. Research Ethics Medical Review Board of El-Minia University has approved the protocol.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2023-09-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of some plasma miRNA profiling in primary ITP and correlation to disease phases and their possible roles in pathogenesis of ITP | 1 May 2022 to 1 September
  Measurement of Micro RNA by qPCR
Explore the cytokines level production of IL-2 in patients with primary ITP at different disease phases and its possible role in pathogenesis of primary ITP | 1 May 2022 to 1 September
  Measurement by ELISA
Explore the cytokines level production of IL-17 in patients with primary ITP at different disease phases and its possible role in pathogenesis of primary ITP | 1 May 2022 to 1 September
  Measurement by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Hend M Moness, professor, Principal Investigator — Faculty Of Medicine, Minya university; Aliaa S Abd EL Fatah, professor, Principal Investigator — Faculty Of Medicine, Minya university; Rasha F Ahmed, professor, Principal Investigator — Faculty of medicine, Minya university
Locations (1):
- Sohag University, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ballantine LE, Ong J, Midgley A, Watson L, Flanagan BF, Beresford MW. The pro-inflammatory potential of T cells in juvenile-onset systemic lupus erythematosus. Pediatr Rheumatol Online J. 2014 Jan 16;12:4. doi: 10.1186/1546-0096-12-4. PMID 24433387
- [Background] Hu Y, Li H, Zhang L, Shan B, Xu X, Li H, Liu X, Xu S, Yu S, Ma D, Peng J, Hou M. Elevated profiles of Th22 cells and correlations with Th17 cells in patients with immune thrombocytopenia. Hum Immunol. 2012 Jun;73(6):629-35. doi: 10.1016/j.humimm.2012.04.015. Epub 2012 Apr 23. PMID 22537755